CLINICAL TRIAL: NCT05274880
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Food Effect on Pharmacokinetic Profiles and Safety of CKD-393 in Healthy Volunteers
Brief Title: Study to Evaluate the Food Effect on Pharmacokinetics Profile and Safety of CKD-393
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A98_06FDI2125
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: CKD-393 administration after a high-fat meal/ Period 2: CKD-393 administration at fasting state
  Interventions: Drug: CKD-393
- Sequence 2 (Experimental): Period 1: CKD-393 administration at fasting state/ Period 2: CKD-393 administration after a high-fat meal
  Interventions: Drug: CKD-393

INTERVENTIONS:
Drug: CKD-393 — PO, QD

SUMMARY:
Study to evaluate the food effect on pharmacokinetic profiles and safety of CKD-393 in healthy volunteers

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover study to evaluate the food effect on pharmacokinetic profiles and safety of CKD-393 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 years old or more and less than 55 years old at screening
2. Individuals who had 17.5 kg/m2 ≤ Body mass index (BMI) < 30.5 kg/m2 and body weight ≥ 55 kg for males and body weight ≥ 50 kg for females

   ☞ BMI = Body weight (kg) / height (m)2
3. Individuals without congenital disease, chronic disease within the last 3 years, or pathological symptoms or signs based on medical examination
4. Individuals who were deemed to be eligible based on the screening tests such as laboratory tests (hematology, chemistry, urinalysis, serology, etc.), vital signs, and 12-lead electrocardiogram
5. Individuals who were willing to participate in the study after being fully informed of the study object and procedures and who signed an informed consent form approved by the institutional review board (IRB) of Korea University Guro Hospital
6. Individuals who agreed to use appropriate contraceptive methods (contraceptive methods other than hormones: condoms, intrauterine devices (IUD, IUS), tubal ligation, cervical cap, diaphragm, etc.) and agreed not to donate sperm during the clinical study and until 1 month after the last administration of investigational product
7. Individuals with the ability and willingness to participate the entire study

Exclusion Criteria:

1. Individuals with medical evidence or clinically significant history of hematological, renal, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic, or immune disease (excluding simple dental histories of dental plaque, impacted tooth, or wisdom tooth, etc.) 1-1) Patients with severe heart failure or who had history of heart failure (New York Heart Association (NYHA) class 1, 2, 3, 4) 1-2) Patients with hepatic failure 1-3) Patients with diabetic ketoacidosis, diabetic coma, or type 1 diabetes mellitus 1-4) Patients with severe infection or trauma, or pre-/post-operative patients 1-5) Patients with edema 1-6) Patients with moderate to severe kidney impairment (eGFR<60 mL/min/1.73 m2) 1-7) Patients who had acute condition that affects renal function such as dehydration, severe infection, cardiovascular collapse (shock), acute myocardial infarction, or sepsis 1-8) Patients who underwent tests using intravenous radioactive iodine contrast (e.g., intravenous urography, intravenous cholangiography, angiography, contrast enhanced computed tomography, etc.) 1-9) Patients with malnutrition, starvation, asthenia, pituitary insufficiency, or adrenal insufficiency 1-10) Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
2. Individuals with a history of gastrointestinal disease (e.g., esophageal achalasia, esophagostenosis, or Crohn's disease) or surgery (excluding simple appendectomy, hernia repair, or tooth extraction) that might affect drug absorption
3. Individuals who had following laboratory test results at screening:

   ☞ ALT or AST > 2x the upper limit of the normal range
4. Individuals who had regular alcohol consumption exceeding 210 g /week within 6 months prior to screening (Beer (5%) 250 mL = 10 g, Soju (20%) 50 mL = 8 g, wine (12%) 125 mL = 12 g)
5. Individuals who smoked 20 cigarettes or more per day within 6 months prior to screening
6. Individuals who had taken any investigational product from other clinical or bioequivalence studies within 6 months prior to the first administration of the investigational product of this study
7. Individuals who had following vital signs at screening:

   ☞ Sitting systolic blood pressure < 90 mmHg or ≥ 160 mmHg or sitting diastolic blood pressure < 60 mmHg or ≥ 100 mmHg
8. Individuals who had serious alcohol or drug abuse history within 1 year prior to the screening
9. Individuals who had taken any drug known as a strong inducer or inhibitor of drug metabolizing enzymes within 30 days prior to the first administration of the investigational product
10. Individuals who had taken prescribed or over-the-counter medicine within 10 days prior to the first administration of the investigational product
11. Individuals who had donated whole blood within 2 months or blood components within 1 month prior to the first administration of the investigational product, or who received transfusion within 1 month prior to the first administration of the investigational product
12. Individuals who had severe acute/chronic medical or mental conditions that might increase the risk caused by study participation or administration of the investigational product or might interfere with the interpretation of study results
13. Individuals with hypersensitivity or history of allergy to the investigational product as well as main ingredients and components of the investigational product (such as tartrazine and sunset yellow FCF)
14. Women who were or might be pregnant and who were breastfeeding
15. Individuals who could not consume the high-fat meal provided during the clinical study
16. Individuals judged by the investigator as inappropriate to participate in the study

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-393 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hours
  AUCt: Area under the curve from dosing to time
Cmax of CKD-393 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hours
  Cmax: Peak plasma drug concentration

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Chung, M.D., Ph.D., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea